CLINICAL TRIAL: NCT05443321
Title: Advancing Health Information Exchange (HIE) During Inter-hospital Transfer (IHT) to Improve Patient Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephanie Mueller, Associate Physician, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P001284
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Infections; Heart Failure; COPD Exacerbation; Asthma; Gastrointestinal Diseases; Cardiac Event; Arrythmia; Renal Failure; Renal Disease; Rheumatic Diseases; Urologic Diseases; Neurologic Disorder; Hematologic Diseases; Oncology Problem; Shock; Critical Illness
MeSH Terms: conditions — Infections; Heart Failure; Asthma; Gastrointestinal Diseases; Cardiovascular Diseases; Arrhythmias, Cardiac; Renal Insufficiency; Kidney Diseases; Rheumatic Diseases; Urologic Diseases; Nervous System Diseases; Hematologic Diseases; Shock; Critical Illness | interventions — Health Information Exchange

STUDY DESIGN:
Intervention Model Description: pre-post interrupted time series analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): The baseline arm will include all included patient transfers from the 3 participating transfer hospitals to the 1 accepting hospital during the 1-year pre-intervention phase. They will not receive any intervention, but rather usual care
- Intervention (Experimental): The intervention arm will include all included patient transfers from the 3 participating transfer hospitals to the 1 accepting hospital during the 1-year intervention phase. They will receive the intervention, which will include utilization of the developed health information exchange platform to transfer clinical information between transferring and accepting hospital. The intervention will not interact directly with the patient, but rather their clinical data.
  Interventions: Other: Health Information Exchange (HIE) platform

INTERVENTIONS:
Other: Health Information Exchange (HIE) platform — An improved health information exchange (HIE) platform will be developed at the start of the study with key stakeholder input. This platform will be implemented for use after baseline data collection, and will allow for improved data exchange between transferring and accepting hospital. We will allow for a 6-month wash-in period prior to intervention data collection.
  Arms: Intervention

SUMMARY:
Sub-optimal transfer of clinical information during inter-hospital transfer (IHT, the transfer of patients between acute care hospitals) is common and can lead to patient harm. To address this problem, the investigators will use key stakeholder input to refine and implement an interoperable health information exchange platform that integrates with the electronic health record and improves the reliability of and access to necessary clinical information in three use cases involving transfer of patients between sending and receiving hospitals with varying levels of affiliation and health record integration. The investigators will assess the effect of this intervention on frequency of medical errors, evaluate the use and usability of this platform from the perspective of those that interact with it, and use these results to develop a dissemination plan to spread implementation and use of this platform across other similar institutions.

DETAILED DESCRIPTION:
The transfer of patients between acute care hospitals (inter-hospital transfer, IHT) is often undertaken to provide patients with needed specialized care that is unavailable at the transferring hospital. IHT occurs regularly, with over 100,000 Medicare patients undergoing IHT annually and with higher frequency among patients with select medical conditions (i.e., acute myocardial infarction), those who are critically ill, and those with multiple chronic conditions (MCC). Although all hospital-based care transitions expose patients to the risks of discontinuity of care, patients who undergo IHT are highly vulnerable to these risks given their illness severity and the fact that IHT involves transfer between providers, settings, and systems of care, thereby lacking potential safe-guards against potential gaps in communication.

The overall goals of this study are to leverage the investigators' extensive research experience in IHT and health information technology innovation, including an in-depth understanding of the essential clinical information required for effective HIE, to design, implement, and rigorously evaluate an intervention to improve HIE during IHT. The investigators propose to implement the intervention in 3 use cases with different levels of integration between sending and receiving hospitals. The platform will use existing data standards to ensure interoperability while also optimizing data visualization and workflow. The investigators will then evaluate the effects of the intervention on medical errors and adverse events, evaluate use and usability of the platform, and conduct a mixed methods evaluation to identify best practices for further refining, disseminating, implementing, and sustaining this intervention across different institutions. To achieve this, the Specific Aims of this study are:

Aim 1: To utilize user-centered design principles and prior knowledge and experience of essential information required during IHT to refine a currently functional inter-operable HIE platform that improves reliability of and access to necessary clinical information during IHT and to implement it in 3 use cases: hospitals within the same health system, hospitals in different systems that share a common EHR, and hospitals in different systems that use different EHRs.

Aim 2: To evaluate the impact of this intervention on clinician-reported medical errors; medical errors attributable to sub-optimal information exchange; adverse events; and other measures of patient safety and workflow, using interrupted time series methodology.

Aim 3: To evaluate the utilization and perceived usability of the HIE platform from the perspective of users who interact with the platform, including clinicians who transfer and accept IHT patients, clinicians at accepting hospitals who admit transferred patients, medical records personnel at transferring hospitals, and access center personnel at accepting hospitals; and identify facilitators and barriers to implementation.

Aim 4: To combine data on use, usability and barriers to implementation from end-users with input from steering committee members to develop a plan for further refinement of the platform and a toolkit for widespread adoption at MGB and dissemination to other similar organizations.

The proposed study will provide a novel, user-centered implementation and evaluation of HIE in order to improve the quality of care and patient outcomes during IHT, an understudied, high-risk care transition impacting a vulnerable patient group. This study includes a purposeful evaluation of IHT between hospitals with different levels of affiliation and EHR integration, in addition to rigorous evaluation of use and usability, and barriers and facilitators of implementation across different institutions to identify best practices for dissemination and implementation. The lessons learned will be used to inform successful and sustained adoption by other health care systems, thus broadly improving care provided to transferred patients.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Transferred from one of the 3 included transferring hospitals (Brigham and Women's Faulkner Hospital, South Shore Hospital, Milford Regional Medical Center)
* Admitted to the general medical, cardiology, oncology, and/or ICU services at Brigham and Women's Hospital

Exclusion Criteria:

* Age < 18 years old
* Transferred from a different acute care hospital than the 3 included hospitals
* Admitted through the ER
* Direct admission from home/clinic
* Admitted to a service other than general medicine, cardiology, oncology or ICU at Brigham and Women's Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Total clinician-reported medical errors | Up to 72 hours after transfer
  Collected via a survey of admitting clinicians 48-72 hours after patient transfer.

SECONDARY OUTCOMES:
Clinician-reported medical errors attributable to poor information exchange | Up to 72 hours after transfer
  Collected via a survey of admitting clinicians 48-72 hours after patient transfer.
Total clinician-reported adverse events | Up to 72 hours after transfer
  Collected via a survey of admitting clinicians 48-72 hours after patient transfer.
Preventable clinician-reported adverse events | Up to 72 hours after transfer
  Collected via a survey of admitting clinicians 48-72 hours after patient transfer.
Ameliorable clinician-reported adverse events | Up to 72 hours after transfer
  Collected via a survey of admitting clinicians 48-72 hours after patient transfer.
Clinician-reported quality of clinical information available | Up to 72 hours after transfer
  Collected via a survey of admitting clinicians 48-72 hours after patient transfer.
Length of stay after transfer | From time-of-day and date of transfer to time-of-day and date of hospital discharge
  Collected from administrative data
Rapid response or ICU transfer within 72-hours of patient transfer | Up to 72-hours after transfer
  Collected from administrative data
Time between acceptance of transfer to patient arrival | Up to 3 days prior to transfer
  Collected from administrative data. From time documented that the patient was accepted for transfer until the time the patient arrives at the transferring hospital
Time between transferred patient arrival and entry of admission orders | Up to 24-hours after transfer
  Collected from administrative data. From time documented that the transferred patient arrived at the accepting hospital until the time that the admission orders were placed

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant data will not be shared with any researchers outside of this study. All data will only be shared in aggregate to any member outside the study team.